CLINICAL TRIAL: NCT04433728
Title: Becoming Adulthood of Phenylketonuric Patients Screened in the Neonatal Period: From 1971 to the Present Day.
Brief Title: Life With Phenylketonuria. Adult Neurological Outcome of PCU Screened Patients From 1971 to 2002.
Acronym: PCU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_28; 2020-A00437-32 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-05-15; First posted 2020-06-16 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Phenylketonurias
Keywords: Becoming neurological in adulthood; Metabolic balance during childhood; Duration and compliance with the low-protein diet
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and dried blood on blotter (dried blood spot) for Phe Rate Whole blood on EDTA for genetics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults Phenylketonuric: Adults patients screened in neonatal period for PKU and treated

SUMMARY:
You were detected during the neonatal period for phenylketonuria and you benefited from the diagnosis of an adapted dietetic care, and this for a variable duration according to the recommendations followed at that time.

The recommendations for the management of phenylketonuria have evolved considerably over time, lengthening the duration, rigor of the diet and target rates. However, few studies have been able to determinate the influence of metabolic balance and pediatric management on fate in adulthood. As you know, the current recommendations are more stringent and prolonged, without taking into account the pediatric data of today's adult patients.

The objective of this study, which is aimed at all adult patients screened and followed by Lille University Hospital, according to the same care methods, allowing a homogeneous monitoring of patients, is to assess the influence of pediatric care (duration of the diet, metabolic balance, compliance) on the future in adulthood. This retrospective and current analysis work could help refine the current recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with classic or atypical phenylketonuria detected in the neonatal period since 1971 in the department of Nord (59) and Pas de Calais (62).
* Patients treated
* Able to receive information
* Patient beneficiary or affiliated to a social security

Exclusion Criteria:

* Patients not screened (born outside French territory) or before 1971.
* Untreated screened patients
* Patients screened for persistent benign hyperphenylalaninaemia not treated with a diet (Phenylalanine level <10 mg / dl or 600 µmol / l without diet to be confirmed)
* Associated confirmed neurological pathology other than a complication of phenylketonuria.
* Refusal to participate in the assessment of Intellectual Quotient in adulthood
* Patient screened, lost to follow-up, found, having moved to another region and not wishing to return to the CHU for follow-up.
* Inability to receive information and or express opposition
* Opposition to participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients screened in Nord Pas de Calais for PKU in the neonatal period since 1971 and treated with a diet and / or drug treatment
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Adult intelligence quotient (IQ) score | Baseline
  Adult intelligence quotient (IQ) score assessed at the last setback in the two groups defined by the duration of the hypoprotidic diet during childhood

SECONDARY OUTCOMES:
The IQ score in adulthood assessed defined by the target Phenylalanine level in one subgroup treated during 8 years. | Baseline, at the last time of decline (= 8 years of low-protein diet)
  The IQ score in adulthood assessed at the last time of decline according to the two subgroups treated during 8 years, defined by the target Phenylalanine level ((2-5 mg/dl versus 8-12 mg/dl)
The IQ score in adulthood assessed according to the length of expanding the Diet (Phe intake) during childhood for children treated during 10 years (target Phe level 2-5 mg/dl) | Baseline,at the last time of decline (= 10 years of low-protein diet)
  The IQ score in adulthood assessed according to length (and degree) of expanding the Diet (increasing Phe intake, during 6 months whatever the Phe levels or longer according the Phe levels) during childhood for children treated during 10 years (xith target Phe level 2-5 mg/dl)
The IQ score in adulthood assessed defined by the metabolic biological parameters in childhood | Baseline
  The IQ score in adulthood assessed at the last time of decline according to the metabolic parameters during childhood
The IQ score in adulthood assessed according to the first phenylalanine level in the target (< 5 mg/dl) | baseline
  The IQ score in adulthood assessed according to the first phenylalanine level in the target (< 5 mg/dl) in the neonatal period

CONTACTS AND LOCATIONS:
Overall Officials: Karine MENTION, MD,PhD, Principal Investigator — University Hospital, Lille